CLINICAL TRIAL: NCT05940597
Title: Pulsed Field Ablation vs Cryoablation In Paroxysmal Atrial Fibrillation
Acronym: FACIL AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC23.0147
Record Dates: First submitted 2023-07-04; First posted 2023-07-11 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation Paroxysmal
MeSH Terms: conditions — Atrial Fibrillation | interventions — Irreversible Electroporation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryoablation arm (Active Comparator): Market approved cryoablation system
  Interventions: Device: Cryoballoon pulmonary vein isolation
- PFA arm (Experimental): Market approved PFA ablation system (Farapulse - Boston Scientific system).
  Interventions: Device: Pulse field ablation

INTERVENTIONS:
Device: Pulse field ablation — ablation of paroxysmal atrial fibrillation by Pulse field ablation
  Arms: PFA arm
Device: Cryoballoon pulmonary vein isolation — ablation of paroxysmal atrial fibrillation by Cryoballoon pulmonary vein isolation
  Arms: Cryoablation arm

SUMMARY:
Cryoballoon pulmonary vein isolation (PVI) has emerged as an alternative to radiofrequency in the treatment of drug-resistant atrial fibrillation (AF). (1) Cryoablation offers potential advantages over radiofrequency, including shorter procedure times, decreased fluoroscopy time, shorter hospital length of stay, and different rates and types of complications. (2) The efficacy over a mean follow-up of one year with cryoablation for AF is comparable to that of radiofrequency ablation in a prospective randomized trial, with a lower major complication rate (3, 4). In recent years, AF cryoablation has established itself as a real alternative to RF ablation, to the point that this ablative source is chosen in one out of five European patients undergoing PV isolation. 70-80% of patients maintain sinus rhythm after a first procedure, showing an efficacy rate equivalent to ablation by RF. It is also comparable to RF when it comes to safety. Phrenic nerve palsy remains the major concern of cryoablation, accounting for 40% of periprocedural complications. A reduction in total procedure time and less dependence on the operator's experience make cryoablation an attractive choice for centres starting an AF ablation program. In conclusion, we do not yet have definitive data to affirm the superiority of one energy source over the other. Generally the choice depends on the availability of the centre and on the experience of the operator.

Pulse field ablation (PFA): Vivek Y. Reddy demonstrates that in patients with paroxysmal atrial fibrillation, PFA rapidly and efficiently isolates PVs with a degree of tissue selectivity and a safety profile(1).PFA can achieve a high degree of durable PV isolation with a comparable efficiency than another techniques (RF or CRYO) at one year follow-up (2) Cryoablation has been a recognised technique for the ablation of atrial fibrillation for many years, with many studies comparing the technique to radiofrequency ablation with equal results. Studies are underway to compare radiofrequency AF ablation versus PFA (BEAT-AF study). A randomized study to compare two methods of cryoablation versus PFA will be necessary to validate the non-inferiority of the technique.

ELIGIBILITY:
Inclusion Criteria:

* The patient is of legal age to participate in the study (age >18 years)
* The patient is eligible for ablation of paroxysmal atrial fibrillation
* The patient or legal representative is able to understand and willing to provide written informed consent to participate in the trial
* The patient is able and willing to return for required follow-up visits and examinations

Exclusion Criteria:

* Previous AF ablation
* Persistent and permanent AF
* The patient is contraindicated or allergic to oral anticoagulation
* The patient or legal representative is enable to understand and willing to provide written informed consent to participate in the trial
* The patient is enable and willing to return for required follow-up visits and examinations
* Pregnant or nursing patient
* Patient in exclusion period of another interventional study,
* Patient under administrative or judicial supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
proportion of subjects experiencing one-year single-procedure clinical success | 12 months
  successful index of AF ablation, absence of atrial arrhythmia recurrence on any type of recording (30 sec by TTM (event monitor), holters, 12-lead ECGs, rhythm strip or other diagnostic ECG documentation), absence of use of class I or III AAD.

SECONDARY OUTCOMES:
Health-related quality of life | 6 and 12 months
  SF-12 questionnaire.
Improvement in AF-specific quality of life | 6 and 12 months
  AFEQT questionnaire
Proportion of patients with death | 12 months
  Death from any causes
Proportion of patients with first hospitalization for cardiovascular causes. | 12 months
  First hospitalization for cardiovascular causes
Proportion of patients with acute complication related to the procedure | during the procedure or one day after
  tamponade, stroke, myocardial infarction, other
Total procedure duration | during the procedure
  Procedure duration in minutes
Total time of fluoroscopy | during the procedure
  Total time of fluoroscopy in minutes
Proportion of patients with embolic events from arrhythmia | 12 months
  Stroke
Long term complications related to the procedure | 12 months
  phrenic palsy, pulmonary vein stenosis, pericarditis, other
Recurrence of atrial fibrillation | 12 months
  Absence of atrial arrhythmia recurrence on any type of recording (30 sec by TTM (event monitor), holters, 12-lead ECGs, rhythm strip or other diagnostic ECG documentation), absence of use of class I or III AAD

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Grenoble Alpes, Grenoble, France